CLINICAL TRIAL: NCT05250999
Title: Comparative Effects of Skin Stretch Sensory Stimuli and Transcutaneous Electrical Nerve Stimulation on Balance in Patients With Diabetic Neuropathy
Brief Title: Skin Stretch Sensory Stimuli and TENS in Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0213 Sobia Younas
Record Dates: First submitted 2022-02-20; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetic Neuropathy; TENS; Kinesiotape; Balance
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Transcutaneous Electric Nerve Stimulation; Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Skin stretch sensory stimuli (Experimental): Skin stretch sensory stimuli along with conventional physiotherapy
  Interventions: Other: Skin stretch sensory stimuli
- Transcutaneous Electrical Nerve Stimulation (Experimental): Transcutaneous electrical nerve stimulation along with conventional physiotherapy
  Interventions: Other: Transcutaneous Electrical nerve stimulation
- Control Group (Active Comparator): Conventional physiotherapy included balance exercises, static exercise and dynamic exercise.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Skin stretch sensory stimuli — Skin stretch sensory stimuli will be exerted by a piece of kinesio tape that as applied above right and left lateral malleolus on posterior leg and on both side of spinous process of second thoracic vertebrae till 15cm below for 24 hours a day, 5 days/ week for 6 weeks along with conventional physiotherapy.
  Arms: Skin stretch sensory stimuli
Other: Transcutaneous Electrical nerve stimulation — TENS will be applied to patient while in sitting position for 30 minutes, twice a week, and for 6 weeks (12 treatment sessions along with conventional physiotherapy). A maximum of 25 m amp electrical stimulation with a biphasic square-wave pattern and a pulse width of 0.5ms in a continuous duty cycle will be used. The intensity of the electrical stimulation will be regulated to the high tolerable level without initiating muscle contractions.
  Arms: Transcutaneous Electrical Nerve Stimulation
Other: Control Group — This program include balance exercises performed twice a week for 6 weeks, which consists of balance, progressive strength, and functional mobility training. Static exercise consists of heel and toe raises, one-legged stance for each limb, weight shifting forward, backward, sideward and diagonally, and turning the head to the left and then to the right keeping the feet together. This exercise comprises two 10-min sessions each, with eyes opened and eyes closed, respectively. Dynamic exercise comprises of walking, step-ups, and bipedal jumps for 10 min. Progressive balance exercises comprises of narrow walking, walking backward, walking sideward, stepping over obstacles, passing, throwing and catching a ball.
  Arms: Control Group

SUMMARY:
The aim of the research was to find and compare the effects of skin stretch sensory stimuli and transcutaneous electrical nerve stimulation (TENS) on balance in diabetic neuropathy. Randomized controlled trial done at District Headquarter hospital Okara. The sample size was 46. The subjects were divided into 3 groups, 15 subjects in skin stretch sensory stimuli group, 15 subjects in TENS group and 16 subjects in control group. Study duration was of 6 month. Sampling technique applied was convenient non-probability sampling. Patients aged range from 45 to 80 years, having moderate peripheral neuropathy, and decrease sensations were included. Tools used in this study were Berg Balance scale and Toronto clinical neuropathy score system. Data was being analyzed through Spss 21.

DETAILED DESCRIPTION:
Literature shows that various studies was done on diabetic patients for pain reduction, increase proprioception, improve muscle function and muscle recruitment by using kinesio tape and transcutaneous electrical nerve stimulation. There is particularly limited literature available on the effects of skin stretch sensory stimuli on balance in DN patients. Therefore, based on the literature study, there is crucial need for studying the effects of skin stretch sensory stimuli and TENS as a treatment approach. Thus, the current study will be an attempt to know the results of skin stretch sensory stimuli and TENS in DN patients.

ELIGIBILITY:
Inclusion Criteria:

* participants age ranged from 45 to 80 years' old
* Both genders.
* patients with moderate peripheral neuropathy 9-11 on Toronto Clinical Neuropathy Scoring system
* HbA1c levels
* peripheral neuropathic pain of >6 months' duration involving the lower extremities
* history of diabetes treated with diet, oral hypoglycemic or insulin therapy
* lower extremity symptoms such as muscle pain, decrease in sensations, Achilles tendon reflex, joint position sense of thumb
* Sensory polyneuropathy because of type 2 diabetic diseases
* Ability to walk household distance without assistance or with the use of assistive device such as cane.

Exclusion Criteria:

* Considerable musculoskeletal deformity such as fracture, amputation, abnormality of ROM.
* Previous history of knee or back surgery
* Lower extremity arthritis that prevents standing
* History of cardiovascular problems such as angina, MI
* Symptomatic postural hypotension
* Foot ulceration.
* Skin problems such as rashes etc.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 6th week
  Berg balance scale is used to quantitively evaluate functional balance in older patients with balance disorders. It is a reliable, valid and sensitive to change scale, that include 14 items, maximum score 56 and required 20-40 minutes for completion. The score showed the patient's ability to control postural balance in which maximum score showed a good functional balance.
Toronto Clinical Neuropathy scoring system | 6th week
  TCNS is a sensitive scoring system to diagnose diabetic neuropathy. The Toronto Clinical Neuropathy Score (TCNS) is for the diagnosis and staging of diabetic neuropathy. The score ranges from a minimum of 0 (no neuropathy) to a maximum of 19 points, and incorporates sensory and motor symptoms, as well lower limb sensory and reflex findings, and symptoms such as numbness, tingling, pain, weakness, ataxia and upper limb symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Aabroo, PPDPT, Principal Investigator — Riphah International University
Locations (1):
- District Head Quarter Hospital, Okara, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No